CLINICAL TRIAL: NCT00847938
Title: Randomized, Controlled, Double-blind, Prospective Study, Comparing Different Doses of Neostigmine at Advanced Decurarization .
Brief Title: Comparision of Different Dose of Neostigmine at Advanced Decurarization
Acronym: NEODEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHD066-08
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Anesthesia
Keywords: neostigmine; neuromuscular blocking agent; train of four; anesthesia
MeSH Terms: interventions — Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): neostigmine 0.04 mg.kg associated with atropine 0.02 mg/kg
  Interventions: Drug: neostigmine
- 2 (Active Comparator): neostigmine 0.02 mg.kg associated with atropine 0.01 mg/kg
  Interventions: Drug: neostigmine
- 3 (Active Comparator): neostigmine 0.1 mg.kg associated with atropine 0.05 mg/kg
  Interventions: Drug: neostigmine
- 4 (No Intervention): no injection of neostigmine

INTERVENTIONS:
Drug: neostigmine — 0.04 mg/kg IV bolus, injection when the of train of four is > or = to 40 %
  Arms: 1
Drug: neostigmine — 0.02 mg/kg IV bolus, injection when the of train of four is > or = to 40 %
  Arms: 2
Drug: neostigmine — 0.01 mg/kg IV bolus, injection when the of train of four is > or = to 40 %
  Arms: 3

SUMMARY:
Neuromuscular blockers (NMB) are currently used in anesthesia. Residual paralysis (RP) due to NMB is responsible for respiratory disorders after extubation. Neuromuscular blockade is monitored by train-of-four (TOF) stimulation at the adductor pollicis. To exclude a RP a mechanomyographic TOF ratio of 0.9 is mandatory. But mecanomyography is not available in clinical routine. Acceleromyography is the most currently monitoring available in daily practice but it has been proved that an acceloromyographic (AMG) TOF ratio of 1.0 is necessary to exclude a RP. The incidence of RP in recovery room is underestimated. So to perform a safe extubation, reversal of the neuromuscular blockade is necessary when an AMG TOF ratio has not reached 1.0. Reversal of neuromuscular blockade is achieved with neostigmine. The recommended dose is 0.04 mg/kg. The administration of neostigmine causes parasympathomimetic effects which has to be reversed with atropine. When neuromuscular blockade is light (AMG TOF ratio of 0.4 which corresponds to the absence of fade at the visual evaluation of the TOF), a low dose of neostigmine might be sufficient with less side effects expected. The goal of the study is to compare the delay between a light neuromuscular block and an AMG TOF ratio of 1.0 for three neostigmine regimens of neostigmine 0.04, 0.02, 0.01 mg/kg with atropine respectively 0.02, 0.01, 0.005 mg/kg and a placebo.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18 years
* informed consent signed
* Patient undergoing any type of scheduled surgery under general anesthesia for which curarization with eventually a maintenance is indicated
* ASA score between I to III

Exclusion Criteria:

* patient > 75 years and < 18 years
* body mass index > 32 mg/m²
* neurology disease, neuromuscular or muscular disease
* peripheral neuropathy
* coronary heart disease
* asthma
* familial history of malign hyperthermia
* difficulty of intubation and ventilation
* full stomach
* known or suspected allergy to one of the study drug
* mecanique obstruction of digestive or urinary tract
* open-angle glaucoma
* patient with risk of urinary retention linked to urethra-prostatic disorder
* concomittant medication with a influence known on neuromuscular (aminosid, anti-convulsif and corticosteroid
* child bearing women or nursing mother
* no affiliation at a social security

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florent Capron, doctor, Principal Investigator — CHD Vendee
Locations (1):
- CHD Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Neostigmine 40 µg/kg: neostigmine 0.04 mg.kg associated with atropine 0.02 mg/kg
  neostigmine: 0.04 mg/kg IV bolus, injection when the of train of four is > or = to 40 %
- Neostigmine 20 µg/kg: neostigmine 0.02 mg.kg associated with atropine 0.01 mg/kg
  neostigmine: 0.02 mg/kg IV bolus, injection when the of train of four is > or = to 40 %
- Neostigmine 10 µg/kg: neostigmine 0.1 mg.kg associated with atropine 0.05 mg/kg
  neostigmine: 0.01 mg/kg IV bolus, injection when the of train of four is > or = to 40 %
- Placebo: no injection of neostigmine
Period: Overall Study
Arm/Group | Neostigmine 40 µg/kg | Neostigmine 20 µg/kg | Neostigmine 10 µg/kg | Placebo
Started | 16 | 15 | 16 | 15
Completed | 16 | 14 | 15 | 15
Not Completed | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neostigmine 40 µg/kg | Neostigmine 20 µg/kg | Neostigmine 10 µg/kg | Placebo | Total
Number analyzed (Participants) | 16 | 14 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (17.6) | 51.9 (18.1) | 60.2 (11.4) | 50.6 (14.8) | 53.3 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 4 | 6 | 22
  Male | 11 | 7 | 11 | 9 | 38
BMI [Mean (Standard Deviation); unit: kg/m²] | 23.9 (3.6) | 25.4 (3.7) | 26.9 (4.0) | 26.9 (3.3) | 25.7 (3.8)
ASA Physical Status Classification System [Count of Participants; unit: Participants] — ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    ASA I | 8 | 6 | 2 | 2 | 18
    ASA II | 8 | 7 | 11 | 13 | 39
    ASA III | 0 | 1 | 2 | 0 | 3
surgery time [Mean (Standard Deviation); unit: minute] | 80.2 (40.4) | 75.8 (32.4) | 84.1 (54.9) | 78.1 (44.3) | 79.6 (43.9)

OUTCOME MEASURES:

1. Primary Outcome: Mesure of the Train-of-four (TOF)
Description: train-of-four monitoring (also known as neuromuscular monitoring), is a technique used during recovery from the application of general anesthesia to objectively determine how well a patient's muscles are able to function, by recording muscle response after nerves electrical stimulation.
Time Frame: from neostigmine injection to TOF ratio = 0.9 and 1.0, evaluated every minute up to 1 hour
Measure: Median (Full Range); unit: minute
Arm/Group | Neostigmine 40 µg/kg | Neostigmine 20 µg/kg | Neostigmine 10 µg/kg | Placebo
Number analyzed (Participants) | 16 | 14 | 15 | 15
minute
  recovery time to TOF ratio of 0.9 | 3.8 [2.3 to 7] | 4.5 [2.5 to 8] | 11.5 [3.8 to 17.5] | 19 [10.5 to 36]
  recovery time to TOF ratio of 1.0 | 5.5 [4 to 11] | 7.8 [3.5 to 11] | 17 [7 to 55] | 26 [20 to 50]

ADVERSE EVENTS:
Arm/Group | Neostigmine 40 µg/kg | Neostigmine 20 µg/kg | Neostigmine 10 µg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes